CLINICAL TRIAL: NCT04837664
Title: Efficacy of Rose Bengal and Curcumin Mediated Photodynamic Therapy in the Treatment of Denture Stomatitis in Patients With Habitual Cigarette Smokers: a Randomized Controlled Clinical Trial
Brief Title: Curcumin; Rose Bengal; Denture Stomatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Labban Nawwaf, Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KingSaudUni
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Candida Albicans Infection; Cigarette Smoking
Keywords: Candida albicans; curcumin; nystatin; photodynamic therapy; rose bengal
MeSH Terms: conditions — Cigarette Smoking | interventions — Curcumin; Rose Bengal; Nystatin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rose Bengal-mediated Photodynamic therapy (Experimental): Participants belonging to the rose bengal mediated photodynamic therapy, their dentures and oral cavity were illuminated using the LED device for 26 minutes (37.5 J/cm2). The photosensitizer rose bengal was sprayed on the palate and dentures for half-hour. To irradiate the palate, the investigator handled the other LED device; the circular platform having LEDs was put within the patient's oral cavity and the illumination of the palate was carried out for 20 minutes (122 J/cm2). The PDT was carried out thrice per week for a half month (6 sessions) in each participant.
  Interventions: Drug: Rose Bengal
- Curcumin-mediated photodynamic therapy (Experimental): Participants belonging to the curcumin mediated photodynamic therapy, their dentures and oral cavity were illuminated using the LED device for 26 minutes (37.5 J/cm2). The photosensitizer curcumin was sprayed on the palate and dentures for half-hour. To irradiate the palate, the investigator handled the other LED device; the circular platform having LEDs was put within the patient's oral cavity and the illumination of the palate was carried out for 20 minutes (122 J/cm2). The PDT was carried out thrice per week for a half month (6 sessions) in each participant.
  Interventions: Drug: Curcumin
- Nystatin therapy (Active Comparator): Participants belonging to the Nystatin group were administered the topical nystatin-based antifungal drug.
  Interventions: Drug: Nystatin

INTERVENTIONS:
Drug: Curcumin — Curcumin was bought from Sigma®, USA, and its solution was freshly prepared by mixing curcumin powder with phosphate-buffered saline.
  Arms: Curcumin-mediated photodynamic therapy
Drug: Rose Bengal — Rose bengal was bought from Sigma®, USA, and its solution was freshly prepared by mixing rose bengal powder with phosphate-buffered saline.
  Arms: Rose Bengal-mediated Photodynamic therapy
Drug: Nystatin — Rinsing with topical nystatin (100,000 UI/mL) suspension for 60 seconds
  Arms: Nystatin therapy

SUMMARY:
Cigarette smoking in conjugation with bad oral hygiene is considered a typical predisposing factor for many oral diseases including denture stomatitis. This study investigated the effect of Rose Bengal (RB)-and Curcumin (CUR)-mediated photodynamic therapy (PDT) in comparison with nystatin therapy in the intervention of denture stomatitis in cigarette smokers. Overall, 45 habitual cigarette smokers aged ~58 years having denture stomatitis were categorized into three groups: Group-I - RB-mediated PDT, Group-II - CUR-mediated PDT, and Group-III - Nystatin therapy. The primary outcome of the interest was: counts of Candida colony from denture surface and palatal mucosa, calculated as CFU/mL, whereas the prevalence of Candida species determined in 3 research groups comprised the secondary outcome. Oral swab specimens were gathered from the denture surfaces and palatal mucosa. All clinical assessments were performed at baseline, 6 weeks, and 12 weeks. C. albicans was the most prevalent yeast identified on both denture surfaces and palatal mucosa, followed by C. tropicalis and C. glabrata. A considerable decrease in the CFU/mL scores were observed in Group-I and Group-II at the end of the interventions and on the 12-week follow-up (p<0.05). Group-I, II, and III demonstrated clinical efficacy rates of 53%, 51%, and 49%, respectively. CUR-and RB-mediated PDT was found to be as effective as topical Nystatin therapy for the intervention of denture stomatitis among cigarette smokers.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria consisted of the following: (1) completely edentulous participants; (2) removable complete denture wearers diagnosed with denture stomatitis (loss of filiform papillae, erythema, and feeling of mucosal burning); and (3) habitual cigarette smokers (individuals smoking at least 1 cigarette per day since ≥3 years).

Exclusion Criteria:

The exclusion criteria consisted of the following: (1) individuals who received steroids, antifungals, or antibiotics over the past 90 days before the initiation of the study; (2) lactating or pregnant women; (3) individuals who had been using the same denture over the past ten years; individuals who underwent cancer treatment (chemotherapy or radiotherapy); (5) patients who are immunocompromised, anemics, or diabetics; (6) habitual alcohol drinkers; and (7) participants who refused to sign the informed consent document.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Candida albican | 12 weeks
  Counts of Candida colony calculated as colony forming unit (CFU)/mL

SECONDARY OUTCOMES:
Candida species | 12 weeks
  Prevalence of other Candida species

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No